CLINICAL TRIAL: NCT00362375
Title: Evaluation of the Healthy Love Workshop, an HIV Prevention Intervention for African American Women by SisterLove, Inc. in Atlanta, GA
Brief Title: Evaluation of the Healthy Love Workshop, an HIV Prevention Intervention for African American Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: SisterLove, Inc. (Other Government)
Responsible Party: Dazon Dixon Diallo, MPH, CEO, SisterLove, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-1927-4768; U65/CCU424514-02 (Other Grant/Funding Number: CDC Cooperative Agreement U65/CCU424514)
Record Dates: First submitted 2006-08-08; First posted 2006-08-10 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-04

CONDITIONS: HIV Infections; Sexually Transmitted Infections
Keywords: Adult; *HIV Infections/pc [Prevention & Control]; Female; Humans; Risk-Taking; Safe Sex; Sexual Behavior; HIV Testing
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Risk-Taking; Safe Sex; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Love Workshop (Experimental): Single-session, small-group HIV prevention intervention
  Interventions: Behavioral: Healthy Love Workshop
- HIV101 (Active Comparator): Single-session, small-group intervention providing facts regarding HIV/AIDS
  Interventions: Behavioral: HIV/AIDS 101 Workshop

INTERVENTIONS:
Behavioral: Healthy Love Workshop — The Healthy Love Workshop is a single-session intervention lasting 3-4 h that is typically delivered to groups of 4-15 women; however, SisterLove facilitators can accommodate larger groups if needed. The intervention is designed to increase consistent use of condoms and other latex barriers, reduce unprotected sex with male partners, and reduce the number of sex partners. HLW also promotes sexual abstinence, HIV testing, and receipt of test results.
  Other Names: Healthy Love Party; Healthy Love
  Arms: Healthy Love Workshop
Behavioral: HIV/AIDS 101 Workshop — The comparison workshop (named HIV101) was also delivered as a single session lasting 2-3 h, to groups of women about the same size and in settings similar to those used for the HLW. The HIV101 workshop consists of an opening, one module containing the same three HIV/STD-related components as the HLW (HIV/AIDS facts, STI facts, and the Look of HIV) and a closing. However, the presentation of this information used a didactic, lecture-style format, as opposed to the interactive approach used to deliver the HLW.
  Other Names: HIV101
  Arms: HIV101

SUMMARY:
The purpose of this program evaluation is to determine whether the Health Love Workshop, a group-level HIV behavioral intervention, reduces HIV-related sex risk behaviors and increases HIV protective behaviors of African American women and women of African descent. The intent of this program is to support an evaluation of the efficacy of the intervention and to provide feedback to the implementing organization to increase intervention effectiveness.

DETAILED DESCRIPTION:
SisterLove, Inc. in Atlanta, Georgia, is evaluating its HIV/AIDS prevention intervention called the Healthy Love Workshop (HLW). The HLW targets African American women and women of African descent who are at risk for HIV infection and transmission. The HLW, which lasts 3 to 4 hours and is delivered during a single session, is a highly interactive workshop that aims to provide a safe environment in which women can learn about: a) the modes of HIV transmission, b) effective strategies for reducing one's risk for contracting or transmitting HIV or other STIs, c) opportunities to develop or enhance skills for self-assessing the risk level of sexual behaviors and the use of safer sex techniques, and d) how to develop an awareness of personal, community and social attitudes, beliefs and norms that influence women's relationships, sexual behavior, and decision-making. SisterLove will identify a minimum of 28 groups of women to participate in the evaluation, which will use a concurrent comparison design with block randomization. These groups will be typical of those that currently receive the HLW, including but not limited to sororities, friendship circles, church groups and other affinity-based groups. Fourteen of the 28 groups will participate in HLW as the intervention group; 14 of the recruited groups will participate in an HIV/AIDS 101 workshop (HIV 101) as the comparison group. Each group will contain about 15 women, thus approximately 420 women will participate in the evaluation. Outcome measures will assess HIV/AIDS knowledge, attitudes towards condom use and HIV testing, condom use intentions, personal HIV/AIDS risk assessment, self-efficacy for taking steps to prevent HIV transmission, consistent condom use, sexual abstinence, and reduction in other sexual risk behaviors. These outcomes will be measured at baseline, and after the intervention at 3- and 6-month follow-ups.

Eligible groups of women were randomly assigned to receive the intervention (15 groups; 161 women) or a comparison workshop (15 groups; 152 women). Behavioral assessments were conducted at baseline and at 3- and 6-month follow-ups. Among sexually active women at the 3-month follow-up, HLW participants were more likely than comparison participants to report having used condoms during vaginal sex with any male partner or with a primary male partner, and to have used condoms at last vaginal, anal or oral sex with any male partner. At the 6-month follow-up, HLW participants were more likely to report condom use at last vaginal, anal or oral sex with any male partner, and having an HIV test and receiving their test results. The study findings suggest that a single-session intervention delivered to pre-existing groups of black women is an efficacious approach to HIV prevention. This study also demonstrates that a CBO can develop and deliver a culturally appropriate, effective HIV prevention intervention for the population it serves and, with adequate resources and technical assistance, rigorously evaluate its intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women of African descent (including African Americans, Caribbean, and African Immigrants)
* Over the age of 18 years

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant
* Do not speak English
* Recent (past 6 months) participation in HIV prevention workshop

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2006-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dazon Dixon Diallo, MPH, Principal Investigator — President/CEO SisterLove, Inc.; Jeffrey H Herbst, PhD, Study Director — Project Officer, Division of HIV/AIDS Prevention, NCHHSTP, CDC; Thomas M Painter, PhD, Study Director — Project Officer, Division of HIV/AIDS Prevention, NCHHSTP, CDC
Locations (1):
- SisterLove, Inc., Atlanta, Georgia, United States

REFERENCES:
- [Result] Diallo DD, Moore TW, Ngalame PM, White LD, Herbst JH, Painter TM. Efficacy of a single-session HIV prevention intervention for black women: a group randomized controlled trial. AIDS Behav. 2010 Jun;14(3):518-29. doi: 10.1007/s10461-010-9672-5. PMID 20135214
- [Derived] Painter TM, Herbst JH, Diallo DD, White LD; Centers for Disease Control and Prevention (CDC). Community-based program to prevent HIV/STD infection among heterosexual black women. MMWR Suppl. 2014 Apr 18;63(1):15-20. PMID 24743662
- See also: SisterLove, Inc. — http://www.sisterlove.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Information about the study was disseminated through print media, public service announcements on local radio stations, electronic communication and informational mailings to local AIDS service organizations, county health departments, medical clinics, and community centers.
Pre-assignment Details: 28 groups did not participate for logistical reasons, including lack of follow-up by group contact (10 groups), failure of women to arrive for the workshop (7 groups), and too few women to meet minimum workshop size (6 groups). Five groups did not participate because of insufficient interest by their members in receiving either workshop.
Groups:
- HIV101: The HIV 101 Workshop is a single-session intervention lasting 3-4 h that is typically delivered to groups of 4-15 women; however, SisterLove facilitators can accommodate larger groups if needed. The intervention is designed to provide factual information regarding HIV/AIDS and sexually transmitted infections.
Period: Overall Study
Arm/Group | Healthy Love Workshop | HIV101
Started | 161 (Number eligible and randomized) | 152 (Number eligible and randomized)
Completed | 121 (Number completed 6-month follow-up assessment) | 117 (Number completed 6-month follow-up assessment)
Not Completed | 40 | 35
Not completed — Lost to Follow-up | 40 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Love Workshop | HIV101 | Total
Number analyzed (Participants) | 161 | 152 | 313
Age Continuous [Mean (Standard Deviation); unit: years] | 29.1 (10.1) | 33.7 (12.7) | 31.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 152 | 313
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 161 | 152 | 313

OUTCOME MEASURES:

1. Primary Outcome: Condom Use During Vaginal Sex With Any Male Partner
Description: Percentage of women who used condoms during vaginal intercourse with any male partner during the past 3 months
Time Frame: Past 3 months
Population: Women who were sexually active at 3-month follow-up and who provided data on outcome measure
Measure: Number; unit: Percent
Arm/Group | Healthy Love Workshop | HIV101
Number analyzed (Participants) | 93 | 94
Percent | 59.3 | 39.6
Statistical Analysis 1: Comparison: HIV101; GEE cluster-adjusted odds ratio; Test type: Superiority or Other; p < 0.05, Generalized Estimating Equation; Odds Ratio (OR) = 2.40, 95% CI 2-sided [1.28 to 4.50]

2. Other Pre Specified Outcome: Sexual Abstinence
Description: The percentage of women who did not engage in vaginal, oral or anal sexual intercourse with male partners
Time Frame: Past 3 months
Population: Based on the number of women who provided valid data at the 3-month follow-up
Measure: Number; unit: Percent
Arm/Group | Healthy Love Workshop | HIV101
Number analyzed (Participants) | 93 | 94
Percent | 36.6 | 43.6
Statistical Analysis 1: Comparison: HIV101; Test type: Superiority or Other; p < 0.05, GEE; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.20 to 1.16]

3. Other Pre Specified Outcome: Unprotected Vaginal Sex With Any Male Partner
Description: The percentage of women who engaged in unprotected vaginal sex (i.e., did not use a condom) with any male partner during the past 3 months
Time Frame: Past 3 months
Population: Based on the number of women who provided valid data at the 3-month follow-up
Measure: Number; unit: Percent
Arm/Group | Healthy Love Workshop | HIV101
Number analyzed (Participants) | 93 | 94
Percent | 37.6 | 36.2
Statistical Analysis 1: Comparison: HIV101; Test type: Superiority or Other; p < 0.05, GEE; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.99 to 1.95]

4. Other Pre Specified Outcome: Number of Male Sex Partners
Description: The number of male sex partners during the past 3 months
Time Frame: Past 3 months
Population: Based on the number of women who provided valid data at the 3-month follow-up
Measure: Mean (Standard Deviation); unit: Number of sex partners
Arm/Group | Healthy Love Workshop | HIV101
Number analyzed (Participants) | 93 | 94
Number of sex partners | 0.70 (0.60) | 0.67 (0.74)
Statistical Analysis 1: Comparison: HIV101; Test type: Superiority or Other; p < 0.05, GEE; GEE incident rate ratio; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.80 to 1.44]

5. Secondary Outcome: HIV Testing and Receipt of Results
Description: Percentage of women who reported testing for HIV infection and received their test results during the past 3 months
Time Frame: Past 3 months
Population: Based on the number of women who provided data at the 3-month follow-up
Measure: Number; unit: Percent
Arm/Group | Healthy Love Workshop | HIV101
Number analyzed (Participants) | 116 | 116
Percent | 20.2 | 16.3
Statistical Analysis 1: Comparison: HIV101; Test type: Superiority or Other; p < 0.05, GEE; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.76 to 2.71]

6. Secondary Outcome: HIV Knowledge
Time Frame: current
Reporting Status: Not Posted

7. Secondary Outcome: Condom Use Self-efficacy
Time Frame: current
Reporting Status: Not Posted

8. Secondary Outcome: Knowledge of HIV Test
Time Frame: current
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Healthy Love Workshop | HIV101
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/152
Other Adverse Events (participants affected / at risk) | 0/161 | 0/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No